CLINICAL TRIAL: NCT05017623
Title: A Multicenter, Open-label, Phase 1 Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of YH003 in Subjects With Advanced Solid Tumors
Brief Title: A Study to Evaluate YH003 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eucure (Beijing) Biopharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YH003003
Record Dates: First submitted 2021-08-12; First posted 2021-08-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention/treatment (Experimental): All subject will receive YH003 intravenously as single agent every three weeks (Q3W) for up to 1 years, until intolerable toxicity, confirmed disease progression, withdrawal of consent, or Investigator decision, whichever comes first.
  Interventions: Drug: YH003

INTERVENTIONS:
Drug: YH003 — All subject will receive YH003 intravenously as single agent every three weeks (Q3W) for up to 1 years, until intolerable toxicity, confirmed disease progression, withdrawal of consent, or Investigator decision, whichever comes first.

SUMMARY:
This is an open-label, dose-escalation study of the study drug YH003 . The study is designed to determine the safety, tolerability and maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of YH003 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1.Subject is willing and able to provide signed and dated informed consent prior to all study-related procedures and is able to comply with all study procedures;
* 2.Patients with histologically or cytologically confirmed solid tumors who have failed standard of care or have no standard of care;
* 3.Male or female, aged ≥ 18 years;
* 4.Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1;
* 5.Have life expectancy of at least 12 weeks based on investigator's judgement;
* 6.Subjects must meet the following laboratory values at the screening visit:

  a）Absolute neutrophil count (ANC) ≥1.5 x 109/L (in absence of growth factor or other support within 2 weeks prior to study entry) ; Platelet count ≥100 x 109/L;Hemoglobin ≥9 g/dL or ≥ 5.6 mmol/L (without growth factor and transfusion support within 14 days prior to study entry . b)Serum creatinine < 1.5 × ULN, calculated creatinine clearance (CrCL) > 50 mL/min (Cockroft-Gault formula) or estimated glomerular filtration rate (GFR) > 50 mL/min; c)Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) and alkaline phosphatase ≤3.0 x ULN; AST or ALT ≤ 5 × ULN if liver metastases are present; d) Serum total bilirubin (TBIL) ≤ 1.5 ULN (for patients with Gilbert's syndrome, TBIL ≤ 3 × ULN); e)International normalized ratio (INR) ≤ 2.0 and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN. Exception: INR 2 to ≤ 3 is acceptable for subjects on Warfarin anticoagulation.
* 7.Women of reproductive potential who are sexually active with a non-sterilized male must consistently use highly effective contraception/birth control between signing of the informed consent and 120 days after the last administration of the study drug.

Exclusion Criteria:

* 1.Previous exposure to TNFR such as anti-CD137, OX40, CD27 and CD357 antibodies.
* 2.Patients with any other malignancy within the past 5 years or currently, except for completely cured non-melanoma skin cancer, carcinoma in situ of the cervix, and ductal carcinoma in situ of the breast;
* 3.Patients with hematological malignancies (such as acute lymphoblastic leukemia, acute myeloid leukemia, myelodysplastic syndrome, multiple myeloma, chronic myelogenous leukemia, non-Hodgkin's lymphoma, Hodgkin's lymphoma, etc.);
* 4.Subjects have received any anticancer therapy or another investigational agent within the shorter of 4 weeks or 5 half-lives before the first dose of the study treatment.Subjects have received Modern traditional Chinese medicine preparations with anti-tumor effect approved by NMPA ≤ 2 weeks prior to first medication.Prior palliative radiotherapy to bone metastases ≤ 2 weeks prior to the first dose of study treatment is acceptable.
* 5.Continuance of toxicities due to prior radiotherapy or chemotherapy agents that have not recovered to ≤ Grade 1 per CTCAE 5.0, except alopecia,≤ Grade 2 sensory neuropathy,lymphopenia, endocrine disease controlled by hormone replacement therapy;.
* 6.Subjects with a history of ≥ Grade 3 immune-related adverse events resulted from previous immunotherapy or treatment discontinuation due to previous immunotherapy.Except hypothyroidism, type 1 diabetes and dermatitis (excluding Steven Johnson syndrome and toxic epidermal necrolysis);
* 7.History of clinically significant sensitivity or allergy to monoclonal antibodies and their excipients or known allergies to antibodies produced from Chinese hamster ovary cells
* 8.Primary central nervous system (CNS) malignancies or symptomatic CNS metastases,except for the following. a) Subjects with asymptomatic brain metastases (No progressive central nervous system symptoms caused by brain metastases, no need for corticosteroids, and lesion size ≤ 1.5 cm);b)Subjects with stable lesions confirmed by imaging examination after local treatment of brain metastases for ≥ 4 weeks, and who discontinued glucocorticoid or anticonvulsant drug treatment 2 weeks before administration of the study drug;
* 9.History of non-infectious pneumonitis or interstitial lung disease that required corticosteroids treatment , except for those caused by radiotherapy, or current interstitial pneumonitis or pneumonitis; or history of other serious lung diseases;
* 10.History of active autoimmune disease, autoimmune disease requiring systemic treatment, or history of autoimmune disease within 2 years prior to the first dose. Exceptions are the following: vitiligo, childhood asthma/idiosyncratic reactions, etc. for which alternative treatments are available;
* 11.Clinically uncontrolled intercurrent illness, including but not limit to uncontrolled diabetes (blood glucose > 250 mg/dl,1 mg/dl=18 mmol/L),uncontrolled hypertension(Systolic blood pressure > 150 mmHg or/and diastolic blood pressure > 100 mmHg),History of hypertension or hypertensive encephalopathy; severe thyroid dysfunction and other serious endocrine diseases or other serious diseases requiring systemic treatment; active infection (such as active pulmonary tuberculosis); active coagulation disorders; other serious diseases requiring systemic treatment;
* 12.Severe cardiovascular disease including symptomatic congestive heart failure (New York Heart Association class III or IV), unstable angina,cardiac arrhythmia, a history of myocardial infarction within 6 months or a history of arterial thromboembolic event and pulmonary embolism within 3 months of the first dose of investigational agent.
* 13.QTc > 470 ms at baseline; Concomitant medications that would prolong the QT interval; Family history of long QT syndrome.
* 14.Subjects must not have active infection of human immunodeficiency virus, hepatitis B, or hepatitis C
* 15. Subjects must not receive concurrent or prior use of an immunosuppressive agent within 4 weeks of the first dose of YH003, with the following exceptions and notes:a)Systemic steroids at physiologic doses (equivalent to dose of oral prednisone 10 mg) are permitted. b)Intranasal, inhaled, topical, intra-articular, and ocular corticosteroids with minimal systemic absorption are permitted.
* 16.Major surgery within 4 weeks prior to study entry and Minor surgery within 2 weeks prior to the first dose of YH003.
* 17.Subjects must not have received a live attenuated vaccine within 28 days before the first dose of YH003, and subjects, if enrolled, should not receive live vaccines during the study or for 180 days after the last dose of YH003.
* 18.Subjects who have had an allogeneic bone marrow transplant or organ transplant.
* 19.Subjects with psychiatric disorder, history of drug abuse, history of drug abuse, or history of alcohol dependence that may affect trial compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | up to 1 year after the last dosing
  The safety will be assessed by monitoring the adverse events (AE) per NCI CTCAE v5.0
Maximum tolerated dose (MTD) and/or Recommended phase 2 dose (RP2D) | up to 1 year after the last dosing
  The MTD and/or RP2D will be determined based on the data of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China